CLINICAL TRIAL: NCT02636062
Title: Predictors of Coronary Artery Calcium Progression in Adults With a Prior Zero Coronary Artery Calcium Score
Status: Withdrawn | Type: Observational
Why Stopped: PI - lack of funding
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dustin M. Thomas, Director, Cardiac CT Imaging and Cardiovascular Research, San Antonio Military Medical Center
Other Study IDs: C.2016.055
Record Dates: First submitted 2015-12-10; First posted 2015-12-21 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease; Endothelial Dysfunction; Atherosclerosis
Keywords: Coronary disease; Coronary artery disease (CAD); Endothelial dysfunction; Coronary artery calcium (CAC)
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biological specimens collected in this study will be used for future testing and evaluation of exploratory systemic biomarkers with respect to prediction of coronary artery disease (CAD) progression and incident development of CAD. Specifically, samples are being collected to investigate pro-fibrotic and pro-inflammatory makers and the effect on CAD development and progression as measured by coronary artery calcification (CAC). DNA samples will be tested for genetic factors and identify trends amongst patients with CAC development, particularly focusing on those with aggressive, multivessel CAC development.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Follow-up CAC > 0: All patients with CAC scores of zero > 5 years previous will be invited to enroll and undergo repeat CAC scanning. This group will include all patients that develop incident CAC.
- Follow-up CAC zero: All patients with CAC scores of zero > 5 years previous will be invited to enroll and undergo repeat CAC scanning. This group will include all patients who continue to have a CAC of zero.

SUMMARY:
This study is a non-randomized prospective cohort study that will define the rate of index atherosclerotic plaque development in adults with a prior coronary artery calcium (CAC) score of 0 given prior CAC zero > 5 years previous. Ancillary testing of serum, whole blood, and endothelial dysfunction will be performed to investigate any detectable systemic processes that predict CAC development.

DETAILED DESCRIPTION:
This study is a non-randomized prospective cohort study that will define the rate of index atherosclerotic plaque development in adults with a prior CAC score of 0 given prior CAC zero > 5 years previous. Study personnel will abstract CAC and coronary computed tomography angiography (CCTA) results on or prior to 31 December 2010 in a single, high-volume military medical center. All patients with CAC scores of zero, irrespective of whether or not this zero CAC was calculated in the presence of a CCTA with non-calcified plaque, will be offered inclusion in the study cohort. Patients will be contacted via telephone and offered study participation. Patients who sign written informed consent will be interviewed to abstract current medical history, medications, exercise practices, and social history. Cardiovascular risk factors of interest will be hypertension, hyperlipidemia, diabetes mellitus, and family history. Patients will then undergo blood draw (complete metabolic panel, complete blood count, lipid panel, serum insulin, high-sensitivity C-reactive protein (CRP), hemoglobin A1c, and thyroid function testing) to screen for undergoing cardiovascular risk factors and to be used as potential risk markers. Additionally, whole blood and serum will be obtained for future investigation to determine new markers of coronary artery disease (CAD) progression and genetic polymorphisms that may predict CAD progression. Patients will also undergo EndoPat testing utilizing an EndoPAT 2000® (digital pulse amplitude tonometry) to assess for endothelial dysfunction. Finally, patients will undergo repeat coronary artery calcium scoring based on standard laboratory protocols based on heart rate and body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Coronary Artery Calcium scoring test graded as 0 Agatston units

Exclusion Criteria:

* Interval development of symptomatic coronary artery disease (defined as prior PCI, CABG, or myocardial infarction) in the time between initial CAC scan and current data review. (These patients will not be enrolled in the trial to undergo repeat CAC testing, but any major cardiovascular events (MACE) will be documented in order to report the 5 year MACE rates amongst CAC zero patients in our population.)
* Pregnant females
* Implantable cardiac pacemaker or defibrillator
* Prior cardiac surgery for valvular heart disease
* Patients with CAC scores ≥ 1
* Patients in atrial fibrillation at the time of CAC acquisition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (> 18 years old) with a prior CAC score of 0 > 5 years ago or more will be contacted to enroll and undergo repeat CAC scanning.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with CAC > 0 | 5 years
  Incident development of any CAC (CAC > 0) between initial scan > 5 years previous and re-scan

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 5 years
  The incidence of major adverse cardiovascular events (defined as death from cardiac cause, myocardial infarction, revascularization of obstructive coronary artery disease, stroke, heart failure, and new onset of atrial fibrillation), in all subjects screened for the study between initial CAC scan demonstrating zero CAC and current study screening.
Per vessel incident CAC | 5 years
  Individual CAC score for each major epicardial coronary vessel in patients with development of incident CAC > 0
Number of patients on statin therapy with incident CAC > 0 compared with statin naïve patients | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dustin M Thomas, MD, Principal Investigator — San Antonio Military Medical Center

IPD SHARING:
Plan to Share IPD: No